CLINICAL TRIAL: NCT02009579
Title: BGOG-cx1/ENGOT-cx1: "Randomized Double-blind Phase II Study Comparing 3-weekly Carboplatin + Paclitaxel With or Without Concomitant and Maintenance Nintedanib (NINTEDANIB) in Advanced or Recurrent Cervical Carcinoma."
Brief Title: ENGOT-cx1/BGOG-cx1: 3 Weekly Carboplatin/Paclitaxel With or Without Nintedanib in Cervix Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Belgian Gynaecological Oncology Group (Other)
Collaborators: Grupo Español de Investigación en Cáncer de Ovario (Other); Mario Negri Gynecologic Oncology group (MaNGO) (Other); Multicenter Italian Trials in Ovarian Cancer (MITO) (Unknown); North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGOG-cx1/ENGOT-cx1
Record Dates: First submitted 2013-10-24; First posted 2013-12-12 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Uterine Cervical Cancer; Paclitaxel; Carboplatin; Nintedanib
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Active Comparator): Nintedanib/vargatef
  Interventions: Drug: Nintedanib
- Comparator arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — Subjects will receive 6 cycles of 3-weekly carboplatin (AUC 5) + paclitaxel (175 mg/m2) and Nintedanib 200 mg BID followed by Nintedanib maintenance until progression or for a total maximum duration of 120 weeks.
  Other Names: Vargatef
  Arms: Experimental arm
Drug: Placebo — Subjects will receive 6 cycles of 3-weekly carboplatin (AUC 5) + paclitaxel (175 mg/m2) and placebo 200 mg BID followed by placebo maintenance until progression or for a total maximum duration of 120 weeks.
  Arms: Comparator arm

SUMMARY:
Indication:

Treatment of subjects with advanced (FIGO stage IVB) or recurrent cervical cancer, prior radiochemotherapy or neo-adjuvant chemotherapy is allowed.

Study design:

This is a phase II randomized, double blind and placebo controlled trial evaluating the efficacy of Nintedanib/placebo in combination with the standard carboplatin and paclitaxel followed by Nintedanib/placebo maintenance in the treatment of patients with advanced or recurrent cervical cancer.

A total of 120 patients will be randomized between the experimental and control arm in a 1:1 ratio. Randomization will be stratified for 1previous chemotherapy for metastatic disease (yes/no) and 2disease status (Stage IVB primary versus recurrent disease).

Experimental arm: Subjects will receive 6 cycles of 3-weekly carboplatin (AUC 5) + paclitaxel (175 mg/m2) and Nintedanib 200 mg BID followed by Nintedanib maintenance until progression or for a total maximum duration of 120 weeks.

Control arm: Subjects will receive 6 cycles of 3-weekly carboplatin (AUC 5) + paclitaxel (175 mg/m2) and placebo 200 mg BID followed by placebo maintenance until progression or for a total maximum duration of 120 weeks.

Subjects without evidence of disease progression after completion or discontinuation of the study treatment will be followed until radiographic disease progression, withdrawal of consent or death.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects more than 18 years of age
* Histologically or cytologically confirmed advanced ([FIGO] stage IVB), or recurrent/persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix will be eligible.
* Prior treatment with angiogenesis inhibitors is allowed
* Up to one prior line of chemotherapy for metastatic cervical cancer is allowed.

  * Treatment of primary disease with concomitant cisplatinum chemotherapy during radiotherapy is allowed and does not count as a line of chemotherapy for metastatic disease.
  * Treatment of primary disease with neoadjuvant chemotherapy before radical local surgery is allowed and does not count as a line of chemotherapy for metastatic disease.
  * Treatment of primary disease with neoadjuvant chemotherapy before radical local surgery followed by adjuvant radiochemotherapy is allowed and does not count as a line of chemotherapy for metastatic disease.
  * Treatment of primary disease with neoadjuvant chemotherapy before radical local surgery followed by adjuvant radiotherapy is allowed and does not count as a line of chemotherapy for metastatic disease.
* Life expectancy at least 3 months.
* ECOG Performance status score of 0 or 1
* At least one measurable lesion according to RECIST 1.1 criteria
* Signed and dated written informed consent prior to admission to the study in accordance with ICH-GCP guidelines and to the local legislation

Exclusion Criteria:

* Known hypersensitivity to the trial drugs or to their excipients (including peanut or soya).
* Brain or leptomeningeal metastases.
* Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels.
* Tumor infiltrating the mucosa of the bowel or bladder, or known fistulas between the tumor and the gastrointestinal or urinary tract.
* Radiographic evidence of cavitary or necrotic tumours
* Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial.
* Therapeutic anticoagulation with drugs requiring INR monitoring (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid <325 mg per day).
* Major injuries within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
* History of clinically significant haemorrhagic or thromboembolic event in the past 6 months.
* Known inherited predisposition to bleeding or thrombosis.
* Significant cardiovascular diseases ( i.e. uncontrolled hypertension, unstable angina within the past 6 months, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion).
* History of a cerebral vascular accident, transient ischemic attack or subarachnoid haemorrhage within the past 6 months.
* Abnormal renal, liver or bone marrow function defined as:

  * Proteinuria CTCAE grade 2 or greater
  * Creatinin > 2 ULN or GFR < 30 ml/min
  * Hepatic function: total bilirubin outside of normal limits; ALT or AST > 1.5 ULN in pts without liver metastasis. For Pts with liver metastases: total bilirubin outside of normal limits, ALT or AST > 2.5 ULN
  * Coagulation parameters: International normalised ratio (INR) > 2, prothrombin time (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional ULN
  * Absolute neutrophil count ( ANC) < 1500/µl, platelets < 100000/µl, haemoglobin < 9.0 g/dl
* Other malignancies within the past 3 years or other malignancy with recurrence in the past 3 years or with high risk of recurrence in the first year. In exception to this rule, the following malignancies may be included: non-melanomatous skin cancer (if adequately treated) , any premalignant (e.g. in situ) carcinoma, or basocellular carcinoma.
* Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy.
* Active or chronic hepatitis C and/or B infection or known HIV infection (based on medical file, only for Italy a mandatory screening test for HIV should be performed for all patients who did not have this test within the last 3 months before the study treatment start).
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug.
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
* Patients of child-bearing potential who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner or sexual abstinence for participating females) during the trial and for at least three months after end of active therapy.
* Pregnancy or breast feeding, female patients must have a negative pregnancy test (β-HCG test in urine or serum) prior to commencing study treatment, if applicable.
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule.
* Active alcohol or drug abuse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2021-01 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 1.5 years after LPI
  Primary objective:
  The purpose of this trial is to determine if chemotherapy (carboplatin/paclitaxel) plus Nintedanib (BIBF 1120) can improve progression free survival compared to chemotherapy (carboplatin/paclitaxel) plus placebo in patients with advanced or recurrent cervical cancer.

SECONDARY OUTCOMES:
Safety and toxicity | 5 years after LPI
  Secondary objectives:
  To evaluate the safety and toxicity reported for of the combination regimen
Overall survival | 5 years after LPI
  To evaluate the response rate according to RECIST 1.1
Patient health status | 5 years after LPI
  To explore the effect of Nintedanib on patient reported health status as measured by EORTC-QOL-Cx 24 and EORTCQLQ-C30 questionnaires
Overall survival | 5 years after LPI
  To evaluate the overall survival

CONTACTS AND LOCATIONS:
Locations (32):
- Belgium (10):
  - CHU Saint-Pierre, Brussels
  - Institut Jules Bordet, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - UZ Antwerpen, Edegem
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - CHR Citadelle, Liège
  - Clinique et maternite St. Elisabeth, Namur
  - Cliniques Universitaires mont godinne, Yvoir
- Germany (6):
  - Charité Med Uni Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Kliniken Essen Mitte, Essen
  - Georg-August University Göttingen, Göttingen
  - Medical University Greifswald, Greifswald
  - University Tübingen, Tübingen
- Italy (11):
  - Centro Riferimento Oncologico, Aviano
  - Spedali Civili, Brescia
  - Azienda Ospedaliera Cannizzaro, Catania
  - National Cancer Institute, Milan
  - Istituto Nazionale Tumori-Pascale Naples, Naples
  - Padova Istituti Oncologico Veneto, Padua
  - University Pisa, Pisa
  - AUSL Reggio Emilia, Reggio Emilia
  - Poloclinico A Gemelli, Rome
  - Mauriziano -Torino, Torino
  - S. Anna Torino, Torino
- Spain (5):
  - Hospital Provincial Reina Sofia, Córdoba
  - H. Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Son Llatzer, Palma Mallorca

REFERENCES:
- See also: BGOG website — http://www.bgog.eu/
- See also: ENGOT website — http://www.esgo.org/engot/Pages/AboutENGOT.aspx